CLINICAL TRIAL: NCT02716402
Title: Cyanotic Congenital Heart Disease: Prevalence of Pulmonary and Cerebral Thrombi-embolic Events
Brief Title: Cyanotic Heart Disease and Thrombosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Annette Schophuus Jensen (Other)
Responsible Party: Sponsor-Investigator, Annette Schophuus Jensen, PhD MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-15012759
Record Dates: First submitted 2016-03-08; First posted 2016-03-23 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Thrombosis
Keywords: Cyanotic congenital heart disease; pulmonary thrombosis; cerebral thrombosis
MeSH Terms: conditions — Thrombosis; Intracranial Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cyanotic congenital heart disease (Other): Patients who previously have been examined with cerebral MRI and V/Q SPECT/CT will be re-examined with cerebral MRI and V/Q SPECT/CT
  Interventions: Radiation: Cerebral MRI and V/Q SPECT/CT

INTERVENTIONS:
Radiation: Cerebral MRI and V/Q SPECT/CT — Cerebral MRI and V/Q SPECT/CT

SUMMARY:
The purpose of the study is to examine previously examined patients with cyanotic congenital heart disease to assess how many of the patients have obtained additional blood clots since they were examined 8 years ago.

DETAILED DESCRIPTION:
Patients with cyanotic congenital heart disease have reduced oxygen content in their blood due to abnormal connection between the heart's right and left sides. The reduced oxygenation of the blood affects several organs of the body and a common complications to the disease is blood clots. Despite the patients are young and do not have typical risk factors, previous studies have shown, that they have a very high prevalence of thrombosis in the lungs and brain.

The reason for the increased prevalence of blood clots is not known. A previous study investigated the prevalence of blood clots systematically in patients with cyanotic congenital heart disease and found that approximately 30-40% of the patients had had a clot in the lung or brain. Thus, the study could not predict, when the patient had had a thrombotic event, and most of the patients did not previously had imaging performed. Therefore the aim of this study is to re-examine previously examined cyanotic patients regardless of previous medical history, to assess how many of the patients have obtained additional blood clots since they were examined 8 years ago.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cyanotic congenital heart disease who have previously participated in the study 'cyanotic congenital heart disease: Hemostatic abnormalities and clinical manifestations' (H-KF-2006-4068).
* Clinically stable

Exclusion Criteria:

* Patients who are not guardians for themselves (not adult).
* Age <18 years.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Pulmonary and cerebral thrombosis | Through study completion, an average of 1 year
  Numbers and locations of cerebral and and pulmonary thrombosis, which will be compared with previous examinations

SECONDARY OUTCOMES:
The total numbers of white matter hyper intensity lessons (WMHL) | Through study completion, an average of 1 year
  The numbers of WMHL will be compared with previous scans.
The size of the white matter hyper intensity lessons (WMHL) | Through study completion, an average of 1 year
  The size of the WMHL will be compared with previous scans.

CONTACTS AND LOCATIONS:
Overall Officials: Annette S Jensen, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Cardiology, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No